CLINICAL TRIAL: NCT02004015
Title: Effect of an Induction Dose of Non Depolarizing Neuro Muscular Blocking Agents (NMBA) on Ultrasound Bowel Peristalsis.
Brief Title: Assessment Study of the Effect of NMBA on Bowel Peristalsis
Acronym: CURARES
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBM_WTR_2012-9
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2015-03

CONDITIONS: Physiopathology
Keywords: Analytical; Diagnostic; Anesthesia; Analgesia
MeSH Terms: conditions — Disease; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atracurium (Experimental): injection of NMBA 0.5 mg/kg milligram(s)/kilogram in Intravenous bolus use
  Interventions: Drug: injection of NMBA
- ROCURONIUM (Experimental): injection of NMBA 0.6 mg/kg milligram(s)/kilogram in Intravenous bolus
  Interventions: Drug: injection of NMBA
- placebo (Placebo Comparator): injection of placebo Injection in Intravenous bolus use
  Interventions: Drug: injection of placebo

INTERVENTIONS:
Drug: injection of placebo — 0.5 mg/kg milligram(s)/kilogram
  Arms: placebo
Drug: injection of NMBA
  Arms: Atracurium; ROCURONIUM

SUMMARY:
Phase III prospective randomised study : curare vs placebo, comparing bowel peristalsis (abdominal echography) in the first minutes of after general anesthesia induction.

Primary End Point: proportion of patients with a score of motion = 0

DETAILED DESCRIPTION:
Primary End Point Proportion of patients with a score of motion = 0

Secondary End Point Time at which thumb adductor twitch measurement disappears (3rd consecutive measure with a twitch at 0) Mean minimal twitch measurement for those patients in who twitch measurement does not disappear Concordance study between twitch measurement and bowel peristalsis XML File Identifier: 1vUwHz2uUXeSc7soLu1cQwRAfcM= Page 15/24 ultrasound score.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* scheduled oro tracheal intubation

Exclusion Criteria:

Counter indication to NMBA:

* predicted difficult airway
* surgical counter indication: facial or laryngeal nerve function monitoring
* allergy to muscle relaxants neuro muscular disease Possible alteration of sensitivity to muscle relaxants due to ongoing medication: ex Valproate or aminoglycoside antibiotics. Predictable alteration of bowel movements or difficult abdominal ultrasound:
* scheduled abdominal surgery
* abdominal surgery in last month
* obesity: body mass index over 30 Full stomach or pregnancy requiring suxamethonium for intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a score of motion = 0 | 10 minutes after NMBA or placebo injection
  Proportion of patients with a score of motion = 0

SECONDARY OUTCOMES:
Time at which thumb adductor twitch measurement disappears | 1 month after injection
  Time at which thumb adductor twitch measurement disappears (3rd consecutive measure with a twitch at 0). Mean minimal twitch measurement for those patients in who twitch measurement does not disappear. Concordance study between twitch measurement and bowel peristalsis

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Taylor, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France